CLINICAL TRIAL: NCT02773355
Title: Timely Detection of Treatment Emergent Serious and Non-serious Adverse Events for Saxenda® in Mexican Patients
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN8022-4210; U1111-1170-6497 (Other: WHO)
Record Dates: First submitted 2016-05-13; First posted 2016-05-16 (Estimated); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Liraglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Saxenda®
  Interventions: Drug: liraglutide 3.0 mg

INTERVENTIONS:
Drug: liraglutide 3.0 mg — Patients will be treated with commercially available Saxenda® prescribed according to routine clinical practice at the discretion of the treating physician.

SUMMARY:
This trial is conducted in North America. The aim is to investigate timely detection of pancreatitis cases as well as cases of suspicion of serious and non-serious adverse reactions possibly or probably related to Saxenda® in Mexican patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol)
* The decision to initiate the treatment with commercially available Saxenda® has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study
* Obese patients (BMI equal to or above 30 kg/m^2) or overweight patients (BMI Equal to or above 27 kg/m^2) with at least one weight related comorbidity according to Saxenda® label text in Mexico
* Age equal or above 18 years at the time of signing informed consent

Exclusion Criteria:

* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Hypersensitivity to Saxenda® or to any of its excipients
* Females of child-bearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (adequate contraceptive measures as required by local law or practice)
* Diagnosis of type 1 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The medical condition investigated in this study is obesity and overweight with one or more weight related comorbidities. The study will aim at observing all patients exposed to Saxenda® during treatment by the 20 participating physicians in Mexico.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2016-05-16 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Frequency of pancreatitis | Year 0-3

SECONDARY OUTCOMES:
Adverse drug reactions (ADR) | Year 0-3

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (3):
- Mexico (3):
  - Novo Nordisk Investigational Site, Monterrey, Nuevo León
  - Novo Nordisk Investigational Site, México, State of Mexico
  - Novo Nordisk Investigational Site, Puebla City

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com